CLINICAL TRIAL: NCT00992381
Title: A Single Centre, Two Treatment, Two Period, Two Sequence, Randomized Crossover Steady-state Relative Bioavailability Study of Naproxen in Two Tablet Formulations Given Twice Daily (PN 400 Tablets Containing 500 mg of Naproxen Plus 20 mg of Esomeprazole Versus Naprosyn® Containing Naproxen 500 mg)
Brief Title: Comparison Study of a New Combination of 2 Marketed Medications (Esomeprazole and Naprosyn) Versus Naprosyn Alone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: POZEN (Industry)
Responsible Party: MCMD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: D1120C00035
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: GI Pain; healthy participants; Safety; bioavailability
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): PN400
  Interventions: Drug: PN400
- 2 (Active Comparator): Naproxen
  Interventions: Drug: Naprosyn

INTERVENTIONS:
Drug: PN400 — 500mg Naproxen and 20mg esomeprazole
  Other Names: VIMOVO™
  Arms: 1
Drug: Naprosyn — 500mg Naproxen
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the absorption of naproxen from the PN 400 combination (Naprosyn and Esomeprazole) tablets is similar to that from the naproxen tablets (Naprosyn®), which are currently sold in Australia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a body weight greater than 50 kg and BMI within the range 18-30(inclusive).
* Subjects must be in good health, as assessed during pre-study medical examination and by review of screening results
* Subjects must understand the procedures involved and agree to participate in the study by giving fully informed, written consent

Exclusion Criteria:

* Significant intercurrent disease of any type, in particular liver, kidney, cardiovascular disease, any form of diabetes or significant gastrointestinal disorder which could affect drug absorption, or any history of gastric or duodenal ulceration.
* Ingestion of any naproxen, omeprazole, esomeprazole or related drugs prior to the recruitment interview, such that these drugs will have been ingested in the 4 weeks prior to the day set for the first Period 1 dose

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-09; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To determine the relative naproxen bioavailability of PN 400 (naproxen 500 mg plus esomeprazole 20 mg) compared to an immediate release Naprosyn® 500 mg tablet | blood samples taken at various time points over 2 treatment periods of 11 days

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic (PK) properties of the naproxen component of PN 400 tablet and immediate release Naprosyn® 500 mg tablet, | Blood samples taken at various time point over 2 periods of 2 days
Compare the adverse event profile of PN 400 with that from Naprosyn® | Adverse event reporting over 2 periods of 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Terry Hurst, Study Director — Q-Pharm Phase one unit; Jo Marjason, Principal Investigator — Q-Pharm Phase one unit
Locations (1):
- Research Site, Brisbane, Queensland, Australia